CLINICAL TRIAL: NCT02995616
Title: Energy Consumption and Cardiorespiratory Load During Robot-Assisted Gait Training in Non-Ambulatory Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Nina Lefeber, Doctoral Researcher, Vrije Universiteit Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LOKOMAT STUDY II
Record Dates: First submitted 2016-12-13; First posted 2016-12-16 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Stroke
Keywords: Robot-Assisted Gait Training; Guidance force; Stroke; Energy Consumption; Cardiorespiratory Load
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lokomat training (Experimental): Patients will be tested in 3 Lokomat training sessions on 3 separate days. During the first session patients will walk in the Lokomat according to their regular therapy settings. During the second and third session patients will walk in the Lokomat with 2 different levels of guidance force (100% guidance force and 60% guidance force).
  Interventions: Device: Regular therapy settings; Device: 100% guidance force; Device: 60% guidance force

INTERVENTIONS:
Device: Regular therapy settings — Patients will walk in the Lokomat according to their regular therapy settings for a minimum of 20 minutes (i.e. minimum tolerable guidance force (GF), minimal tolerable body weight support (BWS) and maximum tolerable walking speed)
Device: 100% guidance force — Patients will walk in the Lokomat with 100% GF for a minimum of 20 minutes (same amount of body weight support and walking speed as in the first session)
Device: 60% guidance force — Patients will walk in the Lokomat with 60% GF for a minimum of 20 minutes (same amount of body weight support and walking speed as in the first session)

SUMMARY:
The aim of this study will be to investigate the energy consumption, cardiorespiratory load and perceived exertion in non-ambulatory subacute stroke patients during a robot-assisted gait training (RAGT) session and to compare the exercise intensity with aerobic training recommendations.

The second aim is to investigate the effect of different levels of guidance force on the energy consumption, cardiorespiratory load and perceived exertion.

DETAILED DESCRIPTION:
STUDY DESIGN. An experimental, 1-group, single-centre trial will be conducted in which stroke patients will perform 2 RAGT sessions: 1) walking in the Lokomat according to regular RAGT settings and 2) walking in the Lokomat with different levels of guidance force (60%, 80% and 100%).

PATIENT RECRUITMENT. We aim to recruit 20 stroke patients in the St. Ursula Rehabilitation Centre in Herk-de-Stad, Belgium.

RESTRICTIONS AND PROHIBITIONS. Patients will be instructed to not consume food, alcohol, caffeine or nicotine at least 3h prior to the intervention. Usual medication intake will be allowed with small amounts of water.

PROCEDURE. Patients will be tested in 3 RAGT sessions on 3 separate days. During the first session patients will walk in the Lokomat according to their regular therapy settings for a minimum of 20 minutes (i.e. minimum tolerable guidance force (GF), minimal tolerable body weight support (BWS) and maximum tolerable walking speed). During the second and third session patients will walk in the Lokomat with 2 different levels of guidance force (once 60% and once 100%) for a minimum 20 minutes each and with the same amount of body weight support and walking speed as in the first session. On a separate day before the intervention, patients will be seated for 10 minutes during which resting values (respiratory gases and heart rate) will be assessed (in order to measure their Resting Metabolic Rate). In addition, informed consent and baseline clinical demographic characteristics will be obtained. At the start of the intervention, a mouth mask, heart rate monitor and gait analysis system will be applied. After a seated resting period of 5 minutes, patients will walk for a minimum of 20 minutes during which respiratory gases and heart rate will be monitored continuously. The Borg rating of perceived exertion will be registered every 3 minutes. The intervention will be terminated early when relative or absolute indications are presented as reported by the American Heart Association or when patients are unable to continue walking. Walking sessions will be controlled for time of day.

RANDOMIZATION. The levels of GF will be randomised..

MATERIALS. A flexible facemask (adult facemask, small/medium, Cortex, Germany), lightweight chest carrying gas analysis system (Metamax 3B, Cortex, Germany) and Bluetooth heart rate belt (Polar H7, Polar Electro, Finland) will be used to measure metabolic and cardiorespiratory parameters. At the start of each measurement, gas (room air and reference gas (17.4% O2 and 5.1% CO2)) and volume (3L syringe) calibrations of the breath-by-breath gas analysis system will be performed in accordance with the manufacturer's instructions.

STATISTICAL ANALYSIS. Statistics will be performed using SPSS (IBM, Chicago, IL). The significance level will be set at 5%. Descriptive statistics will be calculated for baseline patient characteristics. Means and standard deviations will be calculated for continuous variables and frequencies and percentages for categorical variables. To investigate the effect of time and the effect of different levels of guidance force, repeated measures ANOVAs (within subject factors) will be analyzed. In case of significant differences, posthoc analysis will be interpreted. To investigate if the effect of guidance force is related to the patient's baseline level of GF (i.e. GF during regular therapy settings) correlational analysis will be performed and baseline GF will be considered as a covariate.

ELIGIBILITY:
Inclusion Criteria:

* First-ever subacute (≤ 3 months) stroke patients
* Eligible to receive robot-assisted gait training according to local therapists' criteria (i.e. non-ambulatory stroke patients that are able to bear full weight on the hemiplegic leg during a minimum of one gait cycle with manual help allowed to maintain balance)
* Functional Ambulation Category < 3
* Trained in the Lokomat system 2 times prior to the start of the study (i.e. one fitting session and one training session).

Exclusion Criteria:

* > 135 kg and >179 cm
* Unstable cardiovascular conditions
* Musculoskeletal problems (other than stroke) affecting the ability to walk
* Concurrent pulmonary diseases (e.g. asthma)
* Concurrent neurological diseases
* Communicative and/or cognitive problems affecting the ability to comprehend or follow instructions
* Other problems affecting the execution of the intervention (e.g. severe spasticity, contractures or dermatological contra-indications)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Oxygen consumption (VO2) | End 5min resting period; Begin, mid and end of 20min walking period (session 1, 2 and 3)
  Average oxygen consumption (mL/kg/min) at different time frames. Oxygen consumption will be measured continuously (from the beginning of rest till the end of walking). Offline calculations (e.g. averages) will be performed afterwards.
Carbon Dioxide Production (CO2) | End 5min resting period; Begin, mid and end of 20min walking period (session 1, 2 and 3)
  Average carbon dioxide production (mL/kg/min) at different time frames. Carbon dioxide production will be measured continuously (from the beginning of rest till the end of walking). Offline calculations (e.g. averages) will be performed afterwards.
Minute ventilation (VE) | End 5min resting period; Begin, mid and end of 20min walking period (session 1, 2 and 3)
  Average amount of air in- or exhaled (L/min) at different time frames. VE will be measured continuously (from the beginning of rest till the end of the walking session). Offline calculations will be performed afterwards.
Heart rate (HR) | End 5min resting period; Begin, mid and end of 20min walking period (session 1, 2 and 3)
  Average heart rate (beats/min) at different time frames. Heart rate will be measured continuously (from the beginning of rest till the end of the walking session). Offline calculations will be performed afterwards.
Percentage heart rate reserve (%HRR) | Begin, mid and end of 20min walking period (session 1)
  The percentage of the heart rate reserve (i.e. the difference between the person's predicted maximum heart rate and the person's resting heart rate) at different time moments (= heart rate at different times moments divided by predicted heart rate reserve).
Percentage maximal heart rate (%HRmax) | Begin, mid and end of 20min walking period (session 1)
  The percentage of the person's predicted maximal heart rate at different time moments (= heart rate at different times moments divided by predicted maximal heart rate).
Rating of perceived exertion (assessed by the 6-20 Borg scale) (RPE) | End 5min resting period; Begin, mid and end of 20min walking period (session 1, 2 and 3)
  Rating of perceived effort, strain and/or fatigue during walking, pointed on a 15-point Borg scale (6-20) at the end of rest and during walking (every 3 minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Eric Kerckhofs, Prof. Ph.D, Study Chair — Vrije Universiteit Brussel; Eva Swinnen, Prof. Ph.D, Study Director — Vrije Universiteit Brussel; Nina Lefeber, Ph.D student, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- St. Ursula Rehabilitation Centre (Jessa Hospital), Herk-de-Stad, Limburg, Belgium